CLINICAL TRIAL: NCT02688738
Title: Does Preoperative Administration of Oral Doxycycline Decrease the Colonization Rate of Propionibacterium Acnes in the Dermis of the Shoulder?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Model: Parallel | Purpose: Prevention
Other Study IDs: 2016SNam
Record Dates: First submitted 2016-02-11; First posted 2016-02-23 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: Propionibacterium
MeSH Terms: interventions — Doxycycline

ARMS (2):
- Control (No Intervention): Standard of care
- Treatment (Active Comparator): Oral doxycycline
  Interventions: Drug: Doxycycline

INTERVENTIONS:
Drug: Doxycycline
  Arms: Treatment

SUMMARY:
The purpose of this study is to evaluate the ability of oral doxycycline to decrease the colonization of Propionibacterium acnes in the dermis of the shoulder.

ELIGIBILITY:
Inclusion Criteria:

-All male patients (>18 years of age) undergoing shoulder arthroscopy

Exclusion Criteria:

* Female patients
* patients with active acne
* patients who have taken antibiotics in the past month
* doxycycline allergy
* benzoyl peroxide allergy
* clindamycin allergy
* patients with psoriatic/eczematous or other lesions on the shoulder girdle.

Age Groups: Child, Adult, Older Adult
Dates: Start 2015-03; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Quantification of P acnes grown from anaerobic or aerobic culture | within 14 days of surgery